CLINICAL TRIAL: NCT00084201
Title: Cranberry: Interactions With Anti-Infectious Agents
Brief Title: Interactions Between Cranberry Juice and Antibiotics Used to Treat Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R21AT002077-01 (NIH)
Record Dates: First submitted 2004-06-08; First posted 2004-06-09 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-11

CONDITIONS: Urinary Tract Infections
Keywords: Vaccinium macrocarpon
MeSH Terms: conditions — Urinary Tract Infections | interventions — Amoxicillin

INTERVENTIONS:
Drug: Cranberry juice
Drug: Amoxicillin

SUMMARY:
The purpose of study is to determine whether cranberry juice interacts with antibiotics used to treat urinary tract infections (UTIs).

DETAILED DESCRIPTION:
Although evidence of its effectiveness is limited, cranberry juice is widely used to prevent urinary tract infections (UTIs). However, recent studies have shown that cranberry juice may affect the way the body absorbs and metabolizes antibiotics used to treat UTIs. This study will determine whether concurrent cranberry juice administration lowers the urinary concentrations of two commonly used antibiotics, amoxicillin and cefaclor.

This study will involve children being treated for UTIs and adults without UTIs. All of the children will continue their prescribed amoxicillin/cefaclor treatment. After 7 to 10 days of antibiotic treatment, the children will be assigned to receive either cranberry juice for 2 days or no additional treatment. Urine samples will be collected from all child participants before and after the administration of cranberry juice to examine the excretion of the antibiotics.

Adult participants will receive two different doses of amoxicillin, with or without cranberry juice. Blood and urine samples will be collected to evaluate the effect of cranberry juice on the absorption and elimination of amoxicillin.

ELIGIBILITY:
Inclusion Criteria for Children:

* Urinary tract infection (UTI) treated with cefaclor or amoxicillin

Inclusion Criteria for Adults:

* No UTI

Exclusion Criteria:

* Allergies to antibiotics
* Use of medications other than oral contraceptives
* Pregnancy or breast-feeding
* Smoker

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18
Dates: Start 2006-07; Study Completion 2007-06

PRIMARY OUTCOMES:
Drug Elmination

SECONDARY OUTCOMES:
Drug absorption

CONTACTS AND LOCATIONS:
Overall Officials: Gail D Anderson, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States